CLINICAL TRIAL: NCT00778388
Title: Against Pseudomonas Aeruginosa in Healthy Volunteers
Brief Title: Study Assessing Safety and Immunogenicity of IC43 Vaccination Against Pseudomonas Aeruginosa in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IC43-101
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
Keywords: Pseudomonas Aeruginosa
MeSH Terms: conditions — Pseudomonas Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- IC43 50 (Active Comparator): IC43 50 mcg with AI(OH)3
  Interventions: Biological: IC43
- IC43 100 with (Active Comparator): IC43 100 mcg with AI(OH)3
  Interventions: Biological: IC43
- IC43 100 w/o (Active Comparator): IC43 100 mcg w/o AI(OH)3
  Interventions: Biological: IC43
- IC43 200 (Active Comparator): IC43 200 mcg with AI(OH)3
  Interventions: Biological: IC43
- Placebo (Placebo Comparator): Placebo (0,9% NaCl)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: IC43 — The study consists of a screening visit within 14 days before the administration of the investigational medicinal product (IMP), an experimental part of 180 days with seven outpatient visits on days 0, 3, 7, 14, 28, 90 and 180 and with vaccinations on days 0 and 7. IC43 vaccine will be administered intramuscularly during study visit 0 and 7 at three different doses, adjuvanted with Al(OH)3, or in one dose without Al(OH)3. Injection volumes will be 0.5 mL, 1 mL or 2 mL. Placebo will be administered intramuscularly at a dosage of 1 mL.
  Other Names: IC43 Pseudomonas Aeruginosa
  Arms: IC43 100 w/o; IC43 100 with; IC43 200; IC43 50
Drug: Placebo — The study consists of a screening visit within 14 days before the administration of the investigational medicinal product (IMP), an experimental part of 180 days with seven outpatient visits on days 0, 3, 7, 14, 28, 90 and 180 and with vaccinations on days 0 and 7. IC43 vaccine will be administered intramuscularly during study visit 0 and 7 at three different doses, adjuvanted with Al(OH)3, or in one dose without Al(OH)3. Injection volumes will be 0.5 mL, 1 mL or 2 mL. Placebo will be administered intramuscularly at a dosage of 1 mL.
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
The objective is to confirm the optimal dose of IC43 in regard to immunogenicity, safety and tolerability.

DETAILED DESCRIPTION:
The study will be designed as a multi-center, observer-blinded, randomized, placebocontrolled phase 1 study in healthy adult subjects of 18 to 65 years of age. A total of 160 healthy male and female subjects is planned to be enrolled and randomized in five groups receiving different dosages and formulations of IC43 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent obtained prior to study entry
* healthy adults aged between 18 and 65 years
* no clinically relevant pathological findings in any of the investigations at the Screening visit. Minor deviations of laboratory values from the normal range may be accepted, if judged by the investigator to have no clinical relevance
* In female subjects either childbearing potential terminated by surgery or a negative serum pregnancy test during screening and the willingness not to become pregnant during the entire study period by practicing reliable methods of contraception

Exclusion Criteria:

* History of autoimmune diseases and malignancies
* Active or passive vaccination 4 weeks before and during the entire study protocol
* Use of any other investigational or non-registered drug or vaccine in addition to the study vaccine during the study period or within 30 days preceding the first dose of study vaccine
* History of severe hypersensitivity reactions and anaphylaxis
* Known hypersensitivity or allergic reactions to one of the components of the vaccine
* Clinically significant diseases as judged by the investigator
* Immunodeficiency due to immunosuppressive therapy
* A family history of congenital or hereditary immunodeficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
immunogenicity at day 14 | see above
rate of serious adverse events during vaccination period until 6 months after first vaccination | see above
safety laboratory parameters at intervals up to day 180 | see above
systemic and local tolerability at intervals up to day 180 | see above

SECONDARY OUTCOMES:
immunogenicity | see above
measurement of functional antibody induction | see above
measurement of antibody avidity on days 7 and 14 | see above
measurement of anti-histidine antibodies on days 7, 14, 90, and 180 | see above

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Ernsthofer, Mag., Study Director — Valneva Austria GmbH
Locations (3):
- Univ.-Prof. Dr. Bernd Jilma, Vienna, Vienna, Austria
- Germany (2):
  - Dr. Daniel Sehrt, Göttingen, Göttingen
  - Dr. Jutta Harten, Münster, Münster